CLINICAL TRIAL: NCT00841906
Title: Alice PDx User/Validation Extended Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MR-0818-APDxE-MS
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-10

CONDITIONS: Sleep Apnea; Sleep-Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alice PDx with only written instructions (Other): Participants will be asked to follow the Alice PDx user instructions to apply basic leads and sensors and undergo a sleep study in their home. Participants will receive little or no instruction concerning the set up of the Alice PDx device.
  Interventions: Device: Alice PDx with only written instructions
- Alice PDx with written and verbal instructions (Other): Participants will be asked to follow the Alice PDx user instructions to apply basic leads and sensors and undergo a sleep study in their home. Participants will receive little or no instruction concerning the set up of the Alice PDx device.
  Interventions: Device: Alice PDx with written and verbal instructions

INTERVENTIONS:
Device: Alice PDx with only written instructions — Participants will be asked to follow the Alice PDx user instructions to apply basic leads and sensors and undergo a sleep study in their home. Participants will receive little or no instruction concerning the set up of the Alice PDx device. After the Alice PDx home study has proven successful, participants will return to the sleep center to undergo a second sleep study, the Lab Night, in which simultaneous monitoring with the Alice PDx and Alice 5 will be performed.
  Other Names: PDx
  Arms: Alice PDx with only written instructions
Device: Alice PDx with written and verbal instructions — Participants will be provided instruction by a trained sleep professional on the set up of the Alice PDx device. They will then be asked to follow the instructions for the Alice PDx device, if necessary, and undergo a sleep study in their home. After the Alice PDx home study has proven successful, participants will return to the sleep center to undergo a second sleep study, the Lab Night, in which simultaneous monitoring with the Alice PDx and Alice 5 will be performed.
  Other Names: PDx
  Arms: Alice PDx with written and verbal instructions

SUMMARY:
The objective of this study is to test the usability of the Alice PDx device by both the end user (patient/participant) and the sleep technician. Data will be collected via questionnaires regarding the participant's ability to understand the participant user manual under home conditions and the technician's ability to set up the Alice PDx according to the health care provider manual. This study will also compare the physiological data recorded by the Alice PDx to the physiological data recorded by its predicate device the Alice 5 System and validate its equivalence. This will be evaluated by comparing the manual study scores for detected apnea and hypopnea events and on an event by event basis during a standard polysomnography (PSG)/ sleep study. The study will test the ability of the Alice PDx to record good quality data as determined by the Good Study Indicator (GSI) function of the Alice PDx firmware.

The primary hypothesis is that the participant will be able to successfully apply the Alice PDx basic leads following the participant user manual instructions and the sleep technician will be able to successfully apply the advanced leads in preparation for the sleep study. In addition, it will be demonstrated that the Alice PDx is equivalent to the Alice 5 System in its intent to record, display and print physiological data to the clinician/physician in order to aid in the screening/follow-up diagnosis of respiratory sleep disorders.

DETAILED DESCRIPTION:
Alice PDx is a portable, diagnostic recording device. It may be used for obstructive sleep screening as well as follow-up and diagnostic assessment. The device may be used in a sleep lab or clinical setting by trained professionals and it may be used at home by patients as directed by their health care provider. The Alice PDx device is not currently approved by the Food and Drug Administration (FDA).

The Alice PDx device is capable of recording various physiological inputs and storing the data locally on a removable storage card. The device may also be connected directly to a PC (personal computer) running the Alice Sleepware software application. Sleepware can display live or pre-recorded data in a resolution consistent with the computer hardware specifications.

ELIGIBILITY:
Inclusion Criteria:

* Patients must call into a sleep lab or be referred to a sleep lab for a diagnostic polysomnogram
* Able to follow directions
* Able to provide informed consent

Exclusion Criteria:

* Participants requiring supplemental oxygen therapy
* History of having a previous sleep study/polysomnogram performed
* Current positive airway pressure (PAP) users
* Unable or unwilling to perform a polysomnogram

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sukhdev Grover, MD, Principal Investigator — Sleep Center of Greater Pittsburgh; Imran Bajwa, MD, Principal Investigator — Indiana Regional Medical Center Sleep Disorders Center
Locations (2):
- United States (2):
  - Indiana Regional Medical Center Sleep Disorders Center, Indiana, Pennsylvania
  - Sleep Center of Greater Pittsburgh, Monroeville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alice PDx With Only Written Instructions | Alice PDx With Written and Verbal Instructions
Started | 18 | 14
Completed | 16 | 14
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alice PDx With Only Written Instructions | Alice PDx With Written and Verbal Instructions | Total
Number analyzed (Participants) | 18 | 14 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 14 | 32
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.4 (8.8) | 32.6 (6.6) | 34.2 (7.9)
Smoking Status [Number; unit: participants]
  Smokers | 2 | 5 | 7
  Non-Smokers | 16 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: This Study Will Compare the Apnea Hypopnea Index Recorded by the Alice PDx to the Physiological Data Recorded by Its Predicate Device the Alice 5 System and Validate Its Equivalence.
Description: The Apnea-Hypopnea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The AHI detected events of Alice 5 system was compared to the AHI events of the Alice PDx.
Time Frame: Lab Night
Population: All participants that completed the overnight portion of the study were analyzed, they each had an Alice 5 System night and an Alice PDx night.
Measure: Mean (Standard Deviation); unit: events
Groups:
- Alice 5 System; Alice PDx: All participants in the lab night portion of the study will wear an Alice 5 System and an Alice PDx for comparison of the two devices.
Arm/Group | Alice 5 System | Alice PDx
Number analyzed (Participants) | 30 | 30
events | 13.16 (24.69) | 20.24 (24.88)
Statistical Analysis 1: Comparison: Alice 5 System vs Alice PDx; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: This Study Will Compare the Central Apnea Index, Hypopnea Index, Mixed Apnea Index and Obstructive Apnea Index Recorded by the Alice PDx to the Physiological Data Recorded by Its Predicate Device the Alice 5 System and Validate Its Equivalence.
Description: The central apnea index, hypopnea index, mixed apnea index and obstructive apnea indexes are all values that are calculated by determining the type of apneic event (apnea, hypopnea, mixed or obstructive). Each type of event is added up over the night and divided by the number of hours.
  For this analysis each index was compared between both devices.
Time Frame: Lab Night
Population: All participants that completed the overnight portion of the study were analyzed.
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Alice 5 System | Alice PDx
Number analyzed (Participants) | 30 | 30
events/hour
  Central Apnea Index | .18 (.42) | .92 (2.64)
  Hypopnea index | 6.91 (8.33) | 7.15 (4.8)
  Mixed Apnea Index | .12 (.38) | .21 (.52)
  Obstructive Apnea Index | 5.95 (17.54) | 11.97 (21.39)

3. Primary Outcome: This Study Will Compare Different Measurements Recorded by the Alice PDx to the Measurement Data Recorded by Its Predicate Device the Alice 5 System and Validate Its Equivalence.
Description: This study will compare different measurements recorded which include Time in Bed, Stage N1, Stage N2, Stage N3, REM, Sleep Onset Latency, Total Sleep Time, Wake Time in Bed and Wake After Sleep Onset by the Alice PDx to the measurement data recorded by its predicate device the Alice 5 System and validate its equivalence.
Time Frame: Lab Night
Population: All participants that completed the overnight portion of the study were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Alice 5 System | Alice PDx
Number analyzed (Participants) | 30 | 30
minutes
  Time In Bed | 308.61 (385.32) | 178.49 (209.16)
  Time spent in Stage N1 | 5.82 (4.25) | 5.43 (2.73)
  Time spent in Stage N2 | 52.50 (13.51) | 51.05 (9.59)
  Time spent in Stage N3 | 13.03 (8.61) | 13.54 (9.29)
  Time spent in Rapid Eye Movement (REM) | 12.14 (6.88) | 11.74 (5.63)
  Sleep Onset Latency | 16.98 (15.39) | 16.83 (14.35)
  Total Sleep Time | 319.88 (54.55) | 314.93 (58.56)
  Wake Time in Bed | 16.49 (12.24) | 18.23 (12.04)
  Wake After Sleep Onset | 50.57 (46.5) | 55.70 (46.09)

4. Secondary Outcome: The Secondary Objective of This Study is to Compare the Measurements of the Alice PDx When Patients Complete the Set-up of the Device at Home and When Patients Are Set up by a Sleep Technician in the Sleep Laboratory.
Description: The Alice PDx incorporates a unique Good Study Indicator (GSI). The GSI is a predicated on airflow and oximeter signal quality and displays the amount of "good quality data" needed for a study to be complete and valid. The GSI visually displays the amount of good quality data in 25-percent increments on the Alice PDx screen. For purposes of this secondary objective this number was compared from participants who set-up and wore the device at home and those that wore the device in a sleep lab set up by a sleep technician.
Time Frame: Lab Night
Population: 3 participants were not able to provide usable GSI data.
Measure: Mean (Standard Deviation); unit: percentage of average GSI
Groups:
- Alice PDx at Home: All participants set up the Alice PDx at home and in the lab. This is evaluating the Good Study Indicator (GSI) at home.
- Alice PDx in the Lab: All participants set up the Alice PDx at home and in the lab. This is evaluating the Good Study Indicator (GSI) in the lab.
Arm/Group | Alice PDx at Home | Alice PDx in the Lab
Number analyzed (Participants) | 27 | 27
percentage of average GSI | 88.9 (17.4) | 70.3 (31.1)

ADVERSE EVENTS:
Arm/Group | Alice PDx With Only Written Instructions | Alice PDx With Written and Verbal Instructions
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 1/18 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alice PDx With Only Written Instructions (N=18) | Alice PDx With Written and Verbal Instructions (N=14)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No